CLINICAL TRIAL: NCT01706575
Title: A Phase IIb, Open Label, Single Arm, Multicenter Study to Evaluate the Effect of 48-weeks PEG-Interferon Alfa-2a (PEG-IFN) Administration on Serum HBsAg in Chronic Hepatitis B, HBeAg-Negative, Genotype D Patients on Treatment With Nucleos(t)Ide Analogues (NAs), Showing Stable HBV DNA Suppression
Brief Title: A Study of Pegasys (Peginterferon Alfa-2a) Added to Nucleos(t)Ide Analogue Treatment in Participants With HBeAg-Negative Chronic Hepatitis B Genotype D Showing Stable Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Suppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28262; 2012-000080-25 (EudraCT Number)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Pegylated Interferon (Peginterferon) Alfa-2a (Experimental): Participants receiving nucleos(t)ide analogues (NA) therapy with Hepatitis B surface Antigen (HBsAg) decline less than <0.5 log 10 international unit/milliliter (IU/ml) at baseline received peginterferon alfa-2a 180 microgram (mcg), subcutaneously (SC) once weekly for 48 weeks along with their NA therapy.
  Interventions: Drug: Pegylated Interferon (Peginterferon) Alfa-2a; Drug: Nucleos(t)ide Analogues (NA)

INTERVENTIONS:
Drug: Pegylated Interferon (Peginterferon) Alfa-2a — Peginterferon alfa-2a 180 mcg, subcutaneously (SC) once weekly for 48 weeks.
  Other Names: Pegasys
Drug: Nucleos(t)ide Analogues (NA) — Nucleos(t)ide analogues includes adefovir, entecavir, lamivudine or tenofovir.

SUMMARY:
This open-label, single-arm, multicenter study will evaluate the efficacy and safety of adding Pegasys (peginterferon alfa-2a) to nucleos(t)ide analogue (NAs) treatment in participants with HBeAg-negative chronic hepatitis B genotype D showing stable HBV DNA suppression. After a 12-week Lead-in period on treatment with NA, participants with a HBsAg decline <0.5 log10 IU/ml will enter the Add-on period to receive Pegasys 180 mcg subcutaneously weekly for 48 weeks in addition to their current NA treatment. Follow-up will be a further 48 weeks, during which the participants will continue their NA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, 18 - 65 years of age
* Chronic hepatitis B
* Negative for HBeAg
* On monotherapy with any nucleos(t)ide analogue (NA) but telbivudine at enrolment, and HBV DNA persistently below 20 IU/ml for at least 12 months
* HBsAg >100 IU/ml at the beginning of the Lead-in phase, confirmed before addition of Pegasys
* Showing a steady HBsAg kinetic (HBsAg decrease <0.5 log10 IU/ml from Week -12 to start of the Add-on phase)
* Negative pregnancy test for women of childbearing potential
* Women of childbearing potential and fertile males with female partners of childbearing potential must be using reliable contraception during and for 3 months after the Add-on phase

Exclusion Criteria:

* Coinfection with Hepatitis A virus (HAV), Hepatitis C virus (HCV), Hepatitis D virus (HDV), Human Immunodeficiency virus (HIV)
* Evidence of decompensated liver disease (Child-Pugh >/=6)
* History or other evidence of a medical condition associated with chronic liver disease (e.g. hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure)
* Known hypersensitivity to peginterferon alfa-2a
* Pregnant of breastfeeding women
* Evidence of alcohol and/or drug abuse
* History of severe psychiatric disease, especially depression
* History of immunologically mediated disease
* History or evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* History or evidence of severe pulmonary disease associated with functional limitations
* History of severe cardiac disease
* History of severe seizure disorder or current anticonvulsant use
* Evidence of an active or suspected cancer or a history of malignancy (other than basocellular carcinoma or in situ cervical carcinoma) within 5 years prior to study entry
* History of having received any systemic anti-neoplastic (including radiation) or immunomodulatory (including systemic corticosteroids) treatment </= 6 months prior to the first dose or the expectation that such a treatment will be needed at any time during the study
* History or other evidence of severe retinopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Italy (26):
  - A.O. Universitaria Ospedali Riuniti Di Foggia; Malattie Infettive, Foggia, Apulia
  - Foggia, Apulia
  - Nuovo Policlinico; Dipartimento di Malattie Infettive, Napoli, Campania
  - Napoli, Campania
  - UNI DEGLI STUDI - POLICLINICA S. ORSOLA; Dipartimento Malattie dell'Apparato Digerente e Medicina In, Bologna, Emilia-Romagna
  - Bologna, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Medica, Udine, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Policlinico Umberto I Di Roma, Rome, Lazio
  - D.I,M.I.; Cattedra Di Gastroenterologia, Genoa, Liguria
  - Genoa, Liguria
  - Fondazione IRCCS Ospedale Maggiore Policlinico; Gastroenterologia, Milan, Lombardy
  - Milan, Lombardy
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Gastroenterologia, Turin, Piedmont
  - Turin, Piedmont
  - A.O. Universitaria Policlinico Monserrato Di Cagliari; Gastroenterologia, Cagliari, Sardinia
  - Uni Di Cagliari; Dept. Di Scienze Mediche, Cagliari, Sardinia
  - Cagliari, Sardinia
  - Az. Osp. Uni. Ria Policlinico G. Martino; Dept. Di Med. Interna E Terapia Medica - Ii Clinica Medica, Messina, Sicily
  - Messina, Sicily
  - Istituto Di Clinica Medica 1 A; Divisione Di Medicina Generale E Gastroenterologia, Palermo, Sicily
  - Palermo, Sicily
  - Ospedale Cisanello - Az. Osp. Pisana; Unità Operativa Di Gastroenterologia Ed Epatologia, Pisa, Tuscany
  - Pisa, Tuscany
  - Padua, Veneto

REFERENCES:
- [Derived] Lampertico P, Brunetto MR, Craxi A, Gaeta GB, Rizzetto M, Rozzi A, Colombo M; HERMES Study Group. Add-on peginterferon alfa-2a to nucleos(t)ide analogue therapy for Caucasian patients with hepatitis B 'e' antigen-negative chronic hepatitis B genotype D. J Viral Hepat. 2019 Jan;26(1):118-125. doi: 10.1111/jvh.12999. Epub 2018 Dec 11. PMID 30187599

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 76 participants started the study and were included in lead-in period. Out of 76 participants, 70 received study drug.
Period: Overall Study
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Started | 76
Treated | 70
Completed | 64
Not Completed | 12
Not completed — Participant Withdrew Consent | 4
Not completed — Lost to Follow-up | 2
Not completed — Started but not Treated | 6

BASELINE CHARACTERISTICS:
Population: Lead-in participants included all participants enrolled in lead-in period.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.82 (8.46)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent Change From Baseline in Serum Hepatitis B Surface Antigen (HBsAg) Titer at End of the Combination Treatment (Week 48)
Time Frame: Baseline up to Week 48
Population: Per-Protocol Population (PP) included all participants without severe protocol violations, including major inclusion or exclusion criteria violations.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 43
percent change | 59.13 (32.14)

2. Primary Outcome: Efficacy: Percentage of Participants With Serum Hepatitis B Surface Antigen (HBsAg) Decrease >/= 50% From Baseline at End of the Combination Treatment (Week 48)
Description: Participants who stopped pegylated interferon (PEG-IFN) treatment during the add-on phase due to serum HBsAg loss and HBsAg seroconversion were considered as responders.
Time Frame: Baseline and Week 48
Population: PP included all participants without severe protocol violations, including major inclusion or exclusion criteria violations and who were undergoing the Week 48 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 43
percentage of participants | 67.44

3. Secondary Outcome: Efficacy: Change From Baseline in Serum Hepatitis B Surface Antigen (HBsAg) Titer at Week 24, 72 and 96
Description: Change is calculated by HBsAg titer at baseline - HBsAg titer at week of assessments.
Time Frame: Baseline, Week 24, 72 and 96
Population: PP included all participants without severe protocol violations, including major inclusion or exclusion criteria violations. Here, number of participants analyzed signifies those participants who were evaluable for the outcome measure and n signifies the number of participants who were evaluated at specified time points.
Measure: Mean (Standard Deviation); unit: international units per millilitre
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 56
international units per millilitre
  Baseline (n= 56) | 0 (0)
  Change at Week 24 (n= 56) | -546.32 (1215.20)
  Change at Week 72 (n= 55) | -815.69 (1394.89)
  Change at Week 96 (n= 55) | -728.16 (1418.60)

4. Secondary Outcome: Efficacy: Percentage of Participants With HBsAg Decrease >/=1 log10 IU/ml From Baseline to Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 43
percentage of participants | 13.95

5. Secondary Outcome: Efficacy: Number of Participants With Serum HBsAg Loss at Week 12 That Persisted up to Week 96
Description: HBsAg loss is defined as HBsAg less than or equal to (</=) 0.05 IU/ml.
Time Frame: Week 12 up to Week 96
Population: PP included all participants without severe protocol violations, including major inclusion or exclusion criteria violations.
Measure: Number; unit: participants
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 56
participants | 1

6. Secondary Outcome: Efficacy: HBsAg Levels According to Interleukin 28B (IL28B) Genotypes
Time Frame: Baseline and Week 48
Population: Data were not collected, and the outcome measure was not analyzed.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 0

7. Secondary Outcome: Efficacy: HBsAg Levels According to Interferon-Inducible Protein 10 (IP-10) Serum Levels
Time Frame: Baseline and Week 48
Population: Data were not collected, and the outcome measure was not analyzed.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 0

8. Secondary Outcome: Safety: Percentage of Participants With Adverse Events (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to Week 48
Population: Safety population included all participants who received least one dose of the study drug and had at least one post-dose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Number analyzed (Participants) | 69
percentage of participants | 92.75

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Description: Safety Population: Safety population included all participants who received least one dose of the study drug and had at least one post-dose safety assessment.
Arm/Group | Pegylated Interferon (Peginterferon) Alfa-2a
Serious Adverse Events (participants affected / at risk) | 5/69
Other Adverse Events (participants affected / at risk) | 56/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon (Peginterferon) Alfa-2a (N=69)
Papillary thyroid cancer (Endocrine disorders) | 1
Pyrexia (General disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon (Peginterferon) Alfa-2a (N=69)
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 27
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 18
Decreased appetite (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Headache (Nervous system disorders) | 19
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Irritability (Psychiatric disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.